CLINICAL TRIAL: NCT02110459
Title: An Open-label, Non-randomized, Monocenter, Single-dose, Phase I Study to Evaluate Pharmacokinetics and Safety of POL7080 Administered as Single Intravenous Infusion to Subjects With Renal Impairment
Brief Title: Pharmacokinetics and Safety of POL7080 in Patients With Renal Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Polyphor Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: POL7080-005
Record Dates: First submitted 2014-04-08; First posted 2014-04-10 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2016-06

CONDITIONS: Renal Impairment
Keywords: POL7080; Pharmacokinetics
MeSH Terms: conditions — Renal Insufficiency | interventions — murepavadin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Mild renal impairment (Experimental): 3h IV POL7080 infusion
  Interventions: Drug: POL7080
- Moderate renal impairment (Experimental): 3h IV POL7080 infusion
  Interventions: Drug: POL7080
- Severe renal impairment (Experimental): 3h IV POL7080 infusion
  Interventions: Drug: POL7080
- End stage renal disease arm 1 (Experimental): 3h IV POL7080 infusion
  Interventions: Drug: POL7080
- End stage renal disease arm 2 (Experimental): 3h IV POL7080 infusion
  Interventions: Drug: POL7080
- Normal Renal function (Experimental): 3h IV POL7080 infusion
  Interventions: Drug: POL7080

INTERVENTIONS:
Drug: POL7080 — Intravenous infusion

SUMMARY:
To investigate the pharmacokinetics (PK) of POL7080 in subjects with renal function impairment after single intravenous (IV) infusion of POL7080

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who signed informed consent.
2. Male subjects ≥18 and ≤79 years of age; female subjects ≥18 and ≤79 years of age of non-childbearing potential
3. Weight within a BMI range of 19.0-35.0 kg/m2.
4. CLCr according to Cockcroft Gault equation of:

   * 50-80 mL/min (mild renal impairment)
   * 30- <50 mL/min (moderate renal impairment)
   * <30 mL/min (severe renal impairment)
   * subjects receiving dialysis for ≥3 months before dosing (ESRD)
   * >80 mL/min (normal renal function)

Exclusion Criteria:

1. Unwilling or unable to give informed consent.
2. As a result of the medical screening process, the study physician considers the subject unfit for the study.
3. Demonstrating excess in xanthine consumption (more than 5 cups of coffee or equivalent per day).
4. Subjects who smoke more than 10 cigarettes a day.
5. Subjects who consume more than 28 units (males) or more than 21 units (females) of alcohol per week.
6. Any history of hypersensitivity to the IMP.
7. For subjects with renal impairment: No clinically significant change in disease status within at least 1 month prior to study entry, as determined by the investigator.
8. The subject had donated a unit of blood (450 mL) within the 3 months before dosing, or intends to donate in the month after the last scheduled visit.
9. Participation in another clinical study with an investigational drug or device within the last month.
10. Subjects with clinically significant telemetric ECG abnormalities on Day -1
11. Significant allergies requiring intranasal or systemic corticosteroids during any time of the year or history of any anaphylactic reaction.
12. Positive test for human immunodeficiency virus (HIV) antibodies.
13. Acute Hepatitis B or C infection.
14. The subject has tested positive for drugs of abuse at screening.
15. Subjects who have received any prescribed systemic or topical medication within 4 weeks prior to dosing (excluded are those drugs the renally impaired subject is currently taking for treatment of the renal or concomitant disease).
16. Immunocompromised patients (patients after solid organ or bone marrow transplant; patients receiving immunosuppressive treatment).
17. Subjects with known or suspected Pseudomonas infection or colonization (e.g. patients with cystic fibrosis).
18. Subjects with significant liver function abnormalities
19. Subjects with acute myocardial infection or unstable angina pectoris

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2013-04; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
To measure the plasma concentrations of POL7080 | at baseline, 0.5, 1,1.5 and 3 hours after start of infusion, at 1, 2, 3, 4, 5, 6, 8, 12, 24, 48 and 72 hours after end of infusion

SECONDARY OUTCOMES:
Adverse events | Daily assessment up to 7 days from informed consent
  Number of adverse events reported by the patients or observed by the investigator will be recorded. Onset, end date, severity, causal relationship, outcome and measures taken will be summarized. Discontinuations and serious adverse events will be listed and narrative summaries will be provided.
Laboratory abnormalities | Screening, Day -1, Day 2, Day 3, and Day 7
  The number and severity of blood chemistry and hematology findings will be summarized descriptively and compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Atef Halabi, MD, Principal Investigator — CRS Clinical Research Services Kiel GmbH
Locations (1):
- CRS Clinical Research Services Kiel GmbH, Kiel, Germany

REFERENCES:
- [Derived] Dale GE, Halabi A, Petersen-Sylla M, Wach A, Zwingelstein C. Pharmacokinetics, Tolerability, and Safety of Murepavadin, a Novel Antipseudomonal Antibiotic, in Subjects with Mild, Moderate, or Severe Renal Function Impairment. Antimicrob Agents Chemother. 2018 Aug 27;62(9):e00490-18. doi: 10.1128/AAC.00490-18. Print 2018 Sep. PMID 30012756